CLINICAL TRIAL: NCT03308669
Title: Safety, Tolerability, and Pharmacokinetics of Lasmiditan When Co-administered With Topiramate in Healthy Subjects
Brief Title: A Study of Lasmiditan in Healthy Participants When Co-administered With Topiramate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 16925; H8H-MC-LAHT (Other: Eli Lilly and Company)
Record Dates: First submitted 2017-10-09; First posted 2017-10-12 (Actual); Results first posted 2019-11-27 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2018-01

CONDITIONS: Healthy
MeSH Terms: interventions — lasmiditan; Topiramate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Lasmiditan Alone (Experimental): Lasmiditan administered orally, alone
  Interventions: Drug: Lasmiditan
- Placebo Alone (Placebo Comparator): Placebo administered orally, alone
  Interventions: Drug: Placebo
- Topiramate + Lasmiditan (Experimental): Topiramate administered orally, alone, and co-administered with oral lasmiditan
  Interventions: Drug: Lasmiditan; Drug: Topiramate
- Topiramate + Placebo (Experimental): Topiramate administered orally, alone, and co-administered with oral placebo
  Interventions: Drug: Placebo; Drug: Topiramate

INTERVENTIONS:
Drug: Lasmiditan — Administered orally
  Other Names: LY573144
  Arms: Lasmiditan Alone; Topiramate + Lasmiditan
Drug: Placebo — Administered orally
  Arms: Placebo Alone; Topiramate + Placebo
Drug: Topiramate — Administered orally
  Arms: Topiramate + Lasmiditan; Topiramate + Placebo

SUMMARY:
This study will assess the safety, tolerability and blood concentrations of lasmiditan and topiramate together compared to lasmiditan and topiramate separately. Information about any side effects that may occur will be collected.

Participants will be admitted to the Clinical Research Unit (CRU) one day prior to the start of the study and will remain through Day 14.

This study is expected to last approximately 25 days, not including screening. Screening is required within 28 days prior to the start of the study.

ELIGIBILITY:
Inclusion Criteria:

* Are healthy males or females (of non-child bearing potential), as determined by medical history and physical examination
* Have a body mass index of 19.0 to 35.0 kilograms per meter squared (kg/m²) inclusive

Exclusion Criteria:

* Have known allergies to lasmiditan, topiramate, related compounds or any components of the formulation of lasmiditan or topiramate
* Have an abnormal supine blood pressure, defined as systolic blood pressure less than (<) 90 or great (>) 140 millimeters of mercury (mmHg) or diastolic blood pressure <60 or >90 mmHg at screening
* Have known or ongoing psychiatric disorders considered clinically significant by the investigator or demonstrate suicidal ideation on the Columbia Suicide Severity Rating Scale (C-SSRS)
* Have a clinically significant abnormality in the neurological examination
* Have current or a history of orthostatic hypotension (>20-mmHg drop in systolic blood pressure, or >10-mmHg drop in diastolic blood pressure) with or without dizziness and/or syncope at screening or admission to the Clinical Research Unit (CRU) upon repeat testing
* Have an estimated glomerular filtration rate using Modification of Diet in Renal Disease <60 milliliter per minute (mL/min) per 1.73 meter squared (m²)
* Have a history of glaucoma
* Have a history of galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2017-12-02 (Actual); Study Completion 2017-12-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Covance Madison CRU, Madison, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Sequence 1: 50 mg Topiramate + Placebo: Placebo film-coated tablets administered orally once in the morning of Day 1 and once in the morning of Day 14.
  25 milligrams (mg) topiramate administered orally on Day 3, two oral doses separated by approximately 12 hours of a single 25-mg topiramate tablet on Days 4 to 7, and two oral doses of 50 mg (2 × 25-mg tablets) separated by approximately 12 hours on Days 8 to 13.
  Final topiramate dosing (2 25-mg tablets) was co-administered with 1 oral dose of placebo.
- Treatment Sequence 2: 50 mg Topiramate + 200 mg Lasmiditan: 200 mg lasmiditan film-coated tablet administered orally once in the morning of Day 1 and once in the morning of Day 14.
  25 milligrams (mg) topiramate administered orally on Day 3, two oral doses separated by approximately 12 hours of a single 25-mg topiramate tablet on Days 4 to 7, and two oral doses of 50 mg (2 × 25-mg tablets) separated by approximately 12 hours on Days 8 to 13.
  Final topiramate dosing (2 25-mg tablets) was co-administered with 1 oral dose of lasmiditan.
Period: Overall Study
Arm/Group | Treatment Sequence 1: 50 mg Topiramate + Placebo | Treatment Sequence 2: 50 mg Topiramate + 200 mg Lasmiditan
Started | 10 | 20
Received at Least One Dose of Study Drug | 10 | 20
Completed | 10 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- Treatment Sequence 1: 50 mg Topiramate + Placebo: Placebo film-coated tablets administered orally once in the morning of Day 1 and once in the morning of Day 14.
  Two oral doses of 50 mg (2 × 25-mg tablets) separated by approximately 12 hours on Days 8 to 13.
- Treatment Sequence 2: 50 mg Topiramate + 200 mg Lasmiditan: 200 mg lasmiditan film-coated tablet administered orally once in the morning of Day 1 and once in the morning of Day 14.
  Two oral doses of 50 mg (2 × 25-mg tablets) separated by approximately 12 hours on Days 8 to 13.
- Total: Total of all reporting groups
Arm/Group | Treatment Sequence 1: 50 mg Topiramate + Placebo | Treatment Sequence 2: 50 mg Topiramate + 200 mg Lasmiditan | Total
Number analyzed (Participants) | 10 | 20 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.3 (13.3) | 44.0 (13.6) | 44.1 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 10 | 19 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 10 | 19 | 29
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 10 | 11
  White | 9 | 8 | 17
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 20 | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration
Description: A summary of serious and other non-serious adverse events, regardless of causality, is located in the Reported Adverse Events module.
Time Frame: Baseline through Day 24
Population: All participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Placebo administered orally, alone
- 200 mg Lasmiditan: Lasmiditan administered orally, alone
- Topiramate Alone: Topiramate administered orally, alone
- 50 mg Topiramate + 200 mg Lasmiditan: Topiramate administered orally, alone, and co-administered with oral lasmiditan
- 50 mg Topiramate + Placebo: Topiramate administered orally, alone, and co-administered with oral placebo
Arm/Group | Placebo | 200 mg Lasmiditan | Topiramate Alone | 50 mg Topiramate + 200 mg Lasmiditan | 50 mg Topiramate + Placebo
Number analyzed (Participants) | 10 | 20 | 30 | 20 | 10
Participants | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Pharmacokinetics (PK): Maximum Observed Drug Concentration (Cmax) of Topiramate When Administered Alone on Day 13 and When Coadministered With Lasmiditan on Day 14
Description: Pharmacokinetics (PK): Maximum Observed Drug Concentration (Cmax) of Topiramate when administered alone on Day 13 and when coadministered with lasmiditan on Day 14
Time Frame: Day 13 and Day 14: predose,0.5,1,1.5,2,3,4,6,8,12 hours(h)
Population: All participants who received at least one dose of lasmiditan or topiramate and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram/milliliter (ng/mL)
Groups:
- 50 mg Topiramate: 50 mg topiramate administered orally twice-daily on Day 13.
- 50 mg Topiramate + 200 mg Lasmiditan: 50 mg topiramate administered twice-daily Day 14. Single oral Dose of 200 mg lasmiditan on Day 14.
Arm/Group | 50 mg Topiramate | 50 mg Topiramate + 200 mg Lasmiditan
Number analyzed (Participants) | 30 | 20
Nanogram/milliliter (ng/mL) | 4300 (15) | 4190 (16)

3. Secondary Outcome: PK: Maximum Observed Drug Concentration (Cmax) of Lasmiditan When Administered Alone on Day 1 and When Coadministered With Topiramate on Day 14
Description: PK: Maximum Observed Drug Concentration (Cmax) of Lasmiditan When Administered Alone on Day 1 and When Coadministered With Topiramate on Day 14
Time Frame: Day 1 and Day 14: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48 hours
Population: All participants who received at least one dose of lasmiditan or topiramate and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram/milliliter (ng/mL)
Groups:
- 200 mg Lasmiditan: Single Oral Dose of 200 mg lasmiditan alone on Day 1.
- 50 mg Topiramate + 200 mg Lasmiditan: Single oral dose of 200 mg lasmiditan administered on Day 14. 50 mg topiramate administered orally twice-daily on Day 14.
Arm/Group | 200 mg Lasmiditan | 50 mg Topiramate + 200 mg Lasmiditan
Number analyzed (Participants) | 20 | 20
Nanogram/milliliter (ng/mL) | 276 (41) | 301 (35)

4. Secondary Outcome: PK: Area Under the Plasma Concentration Versus Time Curve During One Dosing Interval (AUC [Tau]) of Topiramate When Administered Alone on Day 13 and When Coadministered With Lasmiditan on Day 14
Description: PK: Area Under the Plasma Concentration versus Time Curve During One Dosing Interval (AUC [tau]) of Topiramate When Administered Alone on Day 13 and When Coadministered With Lasmiditan on Day 14
Time Frame: Day 13 and Day 14 - predose,0.5,1,1.5,2,3,4,6,8,12 hours(h)
Population: All participants who received at least one dose of lasmiditan or topiramate and have evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour per milliliter(ng*h/mL)
Arm/Group | 50 mg Topiramate | 50 mg Topiramate + 200 mg Lasmiditan
Number analyzed (Participants) | 30 | 20
nanograms*hour per milliliter(ng*h/mL) | 42600 (15) | 42800 (17)

5. Secondary Outcome: PK: Area Under the Plasma Concentration Versus Time Curve From Zero to Infinity AUC(0-∞) of Lasmiditan When Administered Alone on Day 1 and When Coadministered With Topiramate on Day 14
Description: PK: Area Under the Plasma Concentration versus Time Curve From Zero to Infinity AUC(0-∞) of Lasmiditan When Administered Alone on Day 1 and When Coadministered With Topiramate on Day 14
Time Frame: Day 1 and Day 14: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48 hours
Population: All participants who received at least one dose of lasmiditan or topiramate and have evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour per milliliter(ng*h/mL)
Groups:
- 200 mg Lasmiditan: Single Oral Dose of 200 mg lasmiditan on Day 1.
- 50 mg Topiramate + 200 mg Lasmiditan: Single oral Dose of 200 mg lasmiditan on Day 14. 50 mg topiramate administered twice-daily Day 14.
Arm/Group | 200 mg Lasmiditan | 50 mg Topiramate + 200 mg Lasmiditan
Number analyzed (Participants) | 20 | 20
nanograms*hour per milliliter(ng*h/mL) | 1860 (29) | 2050 (29)

ADVERSE EVENTS:
Time Frame: Up To 24 Days
Description: All participants who received at least one dose of study drug.
Arm/Group | 200 mg Lasmiditan | Placebo | Topiramate Alone | 50 mg Topiramate + 200 mg Lasmiditan | 50 mg Topiramate + Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/10 | 0/30 | 0/20 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/10 | 0/30 | 0/20 | 0/10
Other Adverse Events (participants affected / at risk) | 8/20 | 3/10 | 5/30 | 8/20 | 2/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 200 mg Lasmiditan (N=20) | Placebo (N=10) | Topiramate Alone (N=30) | 50 mg Topiramate + 200 mg Lasmiditan (N=20) | 50 mg Topiramate + Placebo (N=10)
Lip dry (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Scratch (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 7 (7) | 1 (1) | 0 (0) | 5 (5) | 1 (1)
Somnolence (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2) | 3 (3) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Euphoric mood (Psychiatric disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2017-10-20): https://cdn.clinicaltrials.gov/large-docs/69/NCT03308669/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-01): https://cdn.clinicaltrials.gov/large-docs/69/NCT03308669/SAP_001.pdf